CLINICAL TRIAL: NCT03044080
Title: Effects of Repeated Use of Botulinum Neurotoxin Type A (BoNT/A) Free of Complexing Proteins in the Spastic Equinovarus Foot in Stroke Patients: A Randomized Clinical Trial
Brief Title: Effects of Botulinum Neurotoxin Type A (BoNT/A) Free of Complexing Proteins in the Spastic Equinovarus Foot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Esther Duarte, Rehabilitation Research Group Coordinator, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSM/RHB/NR22
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-02

CONDITIONS: Stroke Rehabilitation; Stroke Rehabilitation Spasticity Management
Keywords: Walking Disorder; Stroke; Botulinum Toxin; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IncobotulinumtoxinA (Active Comparator): Injection of 200-300 units of IncobotulinumtoxinA (Xeomin ®)
  Interventions: Drug: IncobotulinumtoxinA
- OnabotulinumtoxinA (Active Comparator): Injection of 200-300 units of onabotulinumtoxiA (Botox®)
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Three consecutive injections of 200-300 units of IncobotulinumtoxinA (Xeomin ®) under ultrasound guidance. The IncobotulinumtoxinA will be distributed according to the individual clinical pattern of spasticity: plantar flexor muscles (triceps sural: gastrocnemius and soleus), tibialis posterior, flexor digitorum longus.
  Arms: IncobotulinumtoxinA
Drug: OnabotulinumtoxinA — ree consecutive injections of 200-300 units of OnabotulinumtoxinA (Botox ®) under ultrasound guidance. The BoNT/A will be distributed according to the individual clinical pattern of spasticity: plantar flexor muscles (triceps sural: gastrocnemius and soleus), tibialis posterior, flexor digitorum longus.
  Arms: OnabotulinumtoxinA

SUMMARY:
Clinical randomized clinical trial to assess the effectiveness on walking speed of repeated use of botulinum neurotoxin type A (BoNT/A)in the post-stroke spastic equinovarus foot in three successive infiltrations at 6-month intervals, checking if the sustainability of the effect is greater in incobotulinumtoxin A (Xeomin®) than in onabotulinumtoxinA (Botox®).

DETAILED DESCRIPTION:
Spasticity is present in 38% of patients at six months after stroke. Equinovarus foot, with or without claw toes and striatal foot, is especially common. There is a weak to moderate evidence in favor of the use of botulinum neurotoxin type A (BoNT/A) in the equinovarus foot, stiff-knee and in other patterns that may interfere with gait ability. Specifically, BoNT/A increases walking speed in stroke patients with spastic equinovarus foot.

Repeated use of BoNT/A may lead to the appearance of neutralizing antibodies, so its effect may decrease over successive infiltrations. Among the differential characteristics of incobotulinumtoxinA (Xeomin®) there is a reduced inactivated botulinum neurotoxin content and the lack of complexing proteins, which would diminish antigenicity and not suppose a decrease of the effect before successive infiltrations.

The objective of this project is to determine the effect on walking speed of repeated use of BoNT/A in post-stroke spinal equinovarus foot in three consecutive injections at 6-month intervals and to investigate whether the sustainability of the effect is greater in incobotulinumtoxinA (Xeomin®) than in onabotulinumtoxinA (Botox®). All patients will receive 200-300 units of BoNT/A (Xeomin ® or Botox ®) that will be distributed according to the individual clinical pattern of spastic equinovarus foot.

ELIGIBILITY:
Inclusion Criteria:

* First-ever Ischemic or haemorrhagic stroke
* Time since stroke onset: >6months
* Hemiparesis with equinovarus foot
* No previous BoNT/A

Exclusion Criteria:

* Non-ambulant patients
* Medical contraindications for BoNT/A use that appear in the product information sheet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in walking speed | Baseline and monthly during 18 months
  Walking speed, expressed in m/s, is assessed in a 10-m corridor

SECONDARY OUTCOMES:
Change in spasticity assessed with the Modified Ashworth Scale | Baseline and monthly during 18 months
  Spasticity assessed with the Modified Ashworth Scale (range 0-5)
Change in walking disability assessed with the Scandinavian Stroke Scale | Baseline and monthly during 18 months
  Walking disability is assessed with the Scandinavian Stroke Scale
Change in functional ambulation ability assessed with the Modified Walking Categories | Baseline and monthly during 18 months
  Functional ambulation ability is assessed with the Modified Walking Categories
Change in step time | Baseline and monthly during 18 months
  Step time (Temporal gait parameter) is expressed in seconds and assessed with instrumented gait analysis
Change in step length | Baseline and monthly during 18 months
  Step length (Spatial gait parameter) is expressed in meters and assessed with instrumented gait analysis

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duarte, PhD, Principal Investigator — Fundació IMIM - Parc de Salut Mar
Locations (1):
- Hospital de l'Esperança, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Background] Watkins CL, Leathley MJ, Gregson JM, Moore AP, Smith TL, Sharma AK. Prevalence of spasticity post stroke. Clin Rehabil. 2002 Aug;16(5):515-22. doi: 10.1191/0269215502cr512oa. PMID 12194622
- [Background] Foley N, Murie-Fernandez M, Speechley M, Salter K, Sequeira K, Teasell R. Does the treatment of spastic equinovarus deformity following stroke with botulinum toxin increase gait velocity? A systematic review and meta-analysis. Eur J Neurol. 2010 Dec;17(12):1419-27. doi: 10.1111/j.1468-1331.2010.03084.x. PMID 20491885
- [Background] Dressler D. Five-year experience with incobotulinumtoxinA (Xeomin((R)) ): the first botulinum toxin drug free of complexing proteins. Eur J Neurol. 2012 Mar;19(3):385-9. doi: 10.1111/j.1468-1331.2011.03559.x. Epub 2011 Oct 28. PMID 22035051